CLINICAL TRIAL: NCT01147250
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate Cardiovascular Outcomes During Treatment With Lixisenatide in Type 2 Diabetic Patients After an Acute Coronary Syndrome
Brief Title: Evaluation of Cardiovascular Outcomes in Patients With Type 2 Diabetes After Acute Coronary Syndrome During Treatment With AVE0010 (Lixisenatide)
Acronym: ELIXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC11319; 2009-012852-26 (EudraCT Number); U1111-1116-5558 (Other: UTN)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to lixisenatide once daily (QD) up to end of treatment.
  Interventions: Drug: Placebo
- Lixisenatide (Experimental): Lixisenatide 10 mcg QD for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010)

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: Sterile aqueous solution; Route of administration: Subcutaneous within 1-hour before breakfast using self-injector pen device (Opticlik®). If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 15 or 10 mcg.
  Other Names: Lyxumia
  Arms: Lixisenatide
Drug: Placebo — Pharmaceutical form: Sterile aqueous solution; Route of administration: Subcutaneous within 1-hour before breakfast.
  Arms: Placebo

SUMMARY:
Primary Objective:

- To demonstrate that lixisenatide can reduce cardiovascular (CV) morbidity and mortality (composite endpoint of CV death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina) compared to placebo in type 2 diabetic participants who recently experienced an acute coronary syndrome (ACS) event.

Secondary Objectives:

To demonstrate that when compared to placebo, lixisenatide can reduce:

* composite endpoint of CV death, non-fatal MI, non-fatal stroke, hospitalization for unstable angina, or hospitalization for heart failure.
* composite endpoint of CV death, non-fatal MI, non-fatal stroke, hospitalization for unstable angina, hospitalization for heart failure, or coronary revascularization procedure.
* urinary albumin excretion (based on the urinary albumin/creatinine ratio).

To assess the safety and tolerability of lixisenatide.

DETAILED DESCRIPTION:
The estimated maximum study duration for the first randomized participant was approximately 204 weeks (± 14 days), with a median follow-up over all participants of approximately 91 weeks, broken down as follows:

* placebo-run-in period: 7 days (+ 3 days)
* double-blind study treatment period: 203 weeks (± 14 days) (with about a 37 months of recruitment period)
* post-treatment follow-up period: 3 days (± 1 day)

All participants were followed from randomization until the end of study, which should occur when the last randomized participant had been followed for approximately 10 months. The actual end date of the study was "event driven" and the study end when there were approximately 844 positively-adjudicated primary cardiovascular outcome events.

ELIGIBILITY:
Inclusion criteria:

* Men and women who experienced a spontaneous ACS event (i.e., ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation MI (NSTEMI) or unstable angina) with a documented elevation above the normal reference range of a cardiac biomarker (Troponin or Creatinine Kinase (CK)-MB) and the clinical presentation consistent with an ACS which lead to admission to an acute care facility, within 180 days following the ACS event and prior to screening.
* Participants with a history of type 2 diabetes (for participants newly diagnosed, diagnosis was based on the World Health Organization (WHO) criteria: i.e., either a fasting venous plasma glucose concentration ≥ 7.0 mmol/L [126 mg/dL] or 2-hour post glucose load venous plasma glucose ≥ 11.1 mmol/L [200 mg/dL], confirmed on 2 occasions) prior to the screening visit.

Exclusion criteria:

* Type 1 diabetes mellitus or history of ketoacidosis within 6 months prior to screening.
* Glycosylated hemoglobin (HbA1c) <5.5 % or >11% measured at screening visit.
* Required to use incretin-based agents (e.g., Glucagon-like peptide -1 (GLP-1) agonists or Dipeptidyl Peptidase-4 (DPP-4) inhibitors) other than the study drug during the double-blind treatment period.
* Participants who had undergone coronary artery bypass graft (CABG) surgery following the qualifying ACS event.
* Participants who had undergone percutaneous coronary intervention (PCI) within 15 days prior to screening.
* Participants with planned revascularization procedure (PCI or CABG) or coronary angiogram within 90 days after screening visit.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease, personal or family history of medullary thyroid cancer (MTC), or genetic conditions that predisposes to MTC (e.g., multiple endocrine neoplasia syndromes).
* Any clinically significant abnormality identified at the time of screening that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study or constrain endpoints assessment such as major systemic diseases.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6068 (Actual)
Dates: Start 2010-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (829):
- United States (200):
  - Investigational Site Number 840415, Birmingham, Alabama
  - Investigational Site Number 840307, Foley, Alabama
  - Investigational Site Number 840692, Mobile, Alabama
  - Investigational Site Number 840037, Mobile, Alabama
  - Investigational Site Number 840210, Mobile, Alabama
  - Investigational Site Number 840326, Muscle Shoals, Alabama
  - Investigational Site Number 840393, Toney, Alabama
  - Investigational Site Number 840656, Mesa, Arizona
  - Investigational Site Number 840506, Phoenix, Arizona
  - Investigational Site Number 840520, Phoenix, Arizona
  - Investigational Site Number 840322, Phoenix, Arizona
  - Investigational Site Number 840250, Tempe, Arizona
  - Investigational Site Number 840042, Tucson, Arizona
  - Investigational Site Number 840303, Hot Springs, Arkansas
  - Investigational Site Number 840184, Jonesboro, Arkansas
  - Investigational Site Number 840361, Little Rock, Arkansas
  - Investigational Site Number 840023, Little Rock, Arkansas
  - Investigational Site Number 840706, Anaheim, California
  - Investigational Site Number 840497, Anaheim, California
  - Investigational Site Number 840667, Downey, California
  - Investigational Site Number 840150, Fresno, California
  - Investigational Site Number 840624, Hawthorne, California
  - Investigational Site Number 840623, Inglewood, California
  - Investigational Site Number 840636, Inglewood, California
  - Investigational Site Number 840455, La Mesa, California
  - Investigational Site Number 840240, Loma Linda, California
  - Investigational Site Number 840262, Long Beach, California
  - Investigational Site Number 840606, Long Beach, California
  - Investigational Site Number 840694, Los Angeles, California
  - Investigational Site Number 840431, Los Angeles, California
  - Investigational Site Number 840135, Los Angeles, California
  - Investigational Site Number 840314, Merced, California
  - Investigational Site Number 840290, Mission Viejo, California
  - Investigational Site Number 840592, National City, California
  - Investigational Site Number 840275, Northridge, California
  - Investigational Site Number 840654, Oakland, California
  - Investigational Site Number 840351, Orange, California
  - Investigational Site Number 840689, Orange, California
  - Investigational Site Number 840582, Pomona, California
  - Investigational Site Number 840346, Port Hueneme, California
  - Investigational Site Number 840466, Roseville, California
  - Investigational Site Number 840575, San Marino, California
  - Investigational Site Number 840131, Santa Ana, California
  - Investigational Site Number 840335, Santa Ana, California
  - Investigational Site Number 840576, Simi Valley, California
  - Investigational Site Number 840414, Sylmar, California
  - Investigational Site Number 840395, Ventura, California
  - Investigational Site Number 840206, Vista, California
  - Investigational Site Number 840480, Westlake Village, California
  - Investigational Site Number 840350, Whittier, California
  - Investigational Site Number 840093, Colorado Springs, Colorado
  - Investigational Site Number 840631, Washington D.C., District of Columbia
  - Investigational Site Number 840044, Washington D.C., District of Columbia
  - Investigational Site Number 840281, Clearwater, Florida
  - Investigational Site Number 840477, Homosassa, Florida
  - Investigational Site Number 840261, Miami, Florida
  - Investigational Site Number 840459, Miami, Florida
  - Investigational Site Number 840432, Oviedo, Florida
  - Investigational Site Number 840318, Panama City, Florida
  - Investigational Site Number 840056, St. Petersburg, Florida
  - Investigational Site Number 840295, Wellington, Florida
  - Investigational Site Number 840066, Atlanta, Georgia
  - Investigational Site Number 840446, Atlanta, Georgia
  - Investigational Site Number 840487, Atlanta, Georgia
  - Investigational Site Number 840578, Blue Ridge, Georgia
  - Investigational Site Number 840534, Columbus, Georgia
  - Investigational Site Number 840447, Duluth, Georgia
  - Investigational Site Number 840499, Duluth, Georgia
  - Investigational Site Number 840536, Idaho Falls, Idaho
  - Investigational Site Number 840413, Pocatello, Idaho
  - Investigational Site Number 840519, Arlington Heights, Illinois
  - Investigational Site Number 840589, Belleville, Illinois
  - Investigational Site Number 840107, Chicago, Illinois
  - Investigational Site Number 840633, Chicago, Illinois
  - Investigational Site Number 840663, Chicago, Illinois
  - Investigational Site Number 840212, Hines, Illinois
  - Investigational Site Number 840345, Joliet, Illinois
  - Investigational Site Number 840681, Peoria, Illinois
  - Investigational Site Number 840360, Elwood, Indiana
  - Investigational Site Number 840676, Gary, Indiana
  - Investigational Site Number 840657, Hammond, Indiana
  - Investigational Site Number 840621, Huntington, Indiana
  - Investigational Site Number 840702, Indianapolis, Indiana
  - Investigational Site Number 840009, Topeka, Kansas
  - Investigational Site Number 840533, Covington, Kentucky
  - Investigational Site Number 840251, Madisonville, Kentucky
  - Investigational Site Number 840168, Owensboro, Kentucky
  - Investigational Site Number 840449, Pikeville, Kentucky
  - Investigational Site Number 840299, Baton Rouge, Louisiana
  - Investigational Site Number 840671, Hammond, Louisiana
  - Investigational Site Number 840470, Metairie, Louisiana
  - Investigational Site Number 840178, Shreveport, Louisiana
  - Investigational Site Number 840043, Annapolis, Maryland
  - Investigational Site Number 840639, Catonsville, Maryland
  - Investigational Site Number 840430, Rockville, Maryland
  - Investigational Site Number 840640, Takoma Park, Maryland
  - Investigational Site Number 840293, Towson, Maryland
  - Investigational Site Number 840019, Alpena, Michigan
  - Investigational Site Number 840352, Buckley, Michigan
  - Investigational Site Number 840555, Chesterfield, Michigan
  - Investigational Site Number 840411, Dearborn, Michigan
  - Investigational Site Number 840205, Detroit, Michigan
  - Investigational Site Number 840581, Flint, Michigan
  - Investigational Site Number 840404, Kalamazoo, Michigan
  - Investigational Site Number 840312, Southfield, Michigan
  - Investigational Site Number 840484, Sterling Heights, Michigan
  - Investigational Site Number 840219, Duluth, Minnesota
  - Investigational Site Number 840199, Eagan, Minnesota
  - Investigational Site Number 840196, Biloxi, Mississippi
  - Investigational Site Number 840445, Kansas City, Missouri
  - Investigational Site Number 840008, Kansas City, Missouri
  - Investigational Site Number 840091, St Louis, Missouri
  - Investigational Site Number 840046, St Louis, Missouri
  - Investigational Site Number 840678, St Louis, Missouri
  - Investigational Site Number 840400, St Louis, Missouri
  - Investigational Site Number 840337, Kalispell, Montana
  - Investigational Site Number 840509, Lincoln, Nebraska
  - Investigational Site Number 840007, Omaha, Nebraska
  - Investigational Site Number 840382, Las Vegas, Nevada
  - Investigational Site Number 840680, Las Vegas, Nevada
  - Investigational Site Number 840217, Las Vegas, Nevada
  - Investigational Site Number 840072, Linden, New Jersey
  - Investigational Site Number 840628, Ridgewood, New Jersey
  - Investigational Site Number 840162, Somerset, New Jersey
  - Investigational Site Number 840285, Albany, New York
  - Investigational Site Number 840585, Jamaica, New York
  - Investigational Site Number 840348, Mineola, New York
  - Investigational Site Number 840119, Northport, New York
  - Investigational Site Number 840696, Rosedale, New York
  - Investigational Site Number 840310, Asheville, North Carolina
  - Investigational Site Number 840454, Calabash, North Carolina
  - Investigational Site Number 840672, Charlotte, North Carolina
  - Investigational Site Number 840152, Charlotte, North Carolina
  - Investigational Site Number 840344, Elizabeth City, North Carolina
  - Investigational Site Number 840328, Greensboro, North Carolina
  - Investigational Site Number 840513, Greensboro, North Carolina
  - Investigational Site Number 840504, Greenville, North Carolina
  - Investigational Site Number 840642, Monroe, North Carolina
  - Investigational Site Number 840481, Raleigh, North Carolina
  - Investigational Site Number 840381, Wilmington, North Carolina
  - Investigational Site Number 840532, Winston-Salem, North Carolina
  - Investigational Site Number 840028, Cincinnati, Ohio
  - Investigational Site Number 840198, Cincinnati, Ohio
  - Investigational Site Number 840543, Columbus, Ohio
  - Investigational Site Number 840456, Dayton, Ohio
  - Investigational Site Number 840368, Marion, Ohio
  - Investigational Site Number 840427, Bend, Oregon
  - Investigational Site Number 840422, Portland, Oregon
  - Investigational Site Number 840511, Portland, Oregon
  - Investigational Site Number 840560, Butler, Pennsylvania
  - Investigational Site Number 840464, Clark Summit, Pennsylvania
  - Investigational Site Number 840401, Pittsburgh, Pennsylvania
  - Investigational Site Number 840266, Providence, Rhode Island
  - Investigational Site Number 840223, Anderson, South Carolina
  - Investigational Site Number 840353, Columbia, South Carolina
  - Investigational Site Number 840529, Greenville, South Carolina
  - Investigational Site Number 840550, Greer, South Carolina
  - Investigational Site Number 840258, Myrtle Beach, South Carolina
  - Investigational Site Number 840309, Taylors, South Carolina
  - Investigational Site Number 840551, Rapid City, South Dakota
  - Investigational Site Number 840524, Bartlett, Tennessee
  - Investigational Site Number 840308, Chattanooga, Tennessee
  - Investigational Site Number 840047, Germantown, Tennessee
  - Investigational Site Number 840313, Jackson, Tennessee
  - Investigational Site Number 840625, Memphis, Tennessee
  - Investigational Site Number 840637, Memphis, Tennessee
  - Investigational Site Number 840096, Nashville, Tennessee
  - Investigational Site Number 840388, Nashville, Tennessee
  - Investigational Site Number 840473, Dallas, Texas
  - Investigational Site Number 840677, Edinburg, Texas
  - Investigational Site Number 840698, El Paso, Texas
  - Investigational Site Number 840439, Fair Oaks Ranch, Texas
  - Investigational Site Number 840164, Houston, Texas
  - Investigational Site Number 840545, Longview, Texas
  - Investigational Site Number 840385, Lubbock, Texas
  - Investigational Site Number 840530, Lubbock, Texas
  - Investigational Site Number 840174, Marshall, Texas
  - Investigational Site Number 840565, Plano, Texas
  - Investigational Site Number 840608, Richmond, Texas
  - Investigational Site Number 840573, San Antonio, Texas
  - Investigational Site Number 840564, Sugarland, Texas
  - Investigational Site Number 840241, Waco, Texas
  - Investigational Site Number 840232, American Fork, Utah
  - Investigational Site Number 840471, Draper, Utah
  - Investigational Site Number 840503, Charlottesville, Virginia
  - Investigational Site Number 840180, Chesapeake, Virginia
  - Investigational Site Number 840465, Chesapeake, Virginia
  - Investigational Site Number 840128, Chesapeake, Virginia
  - Investigational Site Number 840045, Norfolk, Virginia
  - Investigational Site Number 840213, Norfolk, Virginia
  - Investigational Site Number 840001, Richmond, Virginia
  - Investigational Site Number 840286, Roanoke, Virginia
  - Investigational Site Number 840170, Olympia, Washington
  - Investigational Site Number 840094, Spokane, Washington
  - Investigational Site Number 840343, Spokane, Washington
  - Investigational Site Number 840268, Spokane, Washington
  - Investigational Site Number 840061, Tacoma, Washington
  - Investigational Site Number 840613, Fairmount, Wisconsin
  - Investigational Site Number 840121, La Crosse, Wisconsin
  - Investigational Site Number 840493, Milwaukee, Wisconsin
- Argentina (46):
  - Investigational Site Number 032028, Adrogué
  - Investigational Site Number 032030, Bahía Blanca
  - Investigational Site Number 032043, Bahía Blanca
  - Investigational Site Number 032054, Bahía Blanca
  - Investigational Site Number 032066, Caba
  - Investigational Site Number 032049, Caba
  - Investigational Site Number 032056, Caba
  - Investigational Site Number 032003, Caba
  - Investigational Site Number 032017, Capital Federal
  - Investigational Site Number 032009, Capital Federal
  - Investigational Site Number 032050, Cipolletti
  - Investigational Site Number 032052, Ciudad Autonoma de Bs.As
  - Investigational Site Number 032020, Coronel Suárez
  - Investigational Site Number 032004, Corrientes
  - Investigational Site Number 032018, Corrientes
  - Investigational Site Number 032015, Córdoba
  - Investigational Site Number 032011, Córdoba
  - Investigational Site Number 032022, Córdoba
  - Investigational Site Number 032037, Córdoba
  - Investigational Site Number 032005, Godoy Cruz
  - Investigational Site Number 032042, Haedo
  - Investigational Site Number 032019, Junín
  - Investigational Site Number 032063, La Plata
  - Investigational Site Number 032040, Lanús
  - Investigational Site Number 032036, Mar del Plata
  - Investigational Site Number 032039, Mar del Plata
  - Investigational Site Number 032058, Mendoza
  - Investigational Site Number 032038, Morón
  - Investigational Site Number 032002, Paraná
  - Investigational Site Number 032023, Qilmes
  - Investigational Site Number 032047, Rafaela
  - Investigational Site Number 032024, Ramos Mejía
  - Investigational Site Number 032006, Resistencia
  - Investigational Site Number 032012, Rosario
  - Investigational Site Number 032027, Rosario
  - Investigational Site Number 032055, Salta
  - Investigational Site Number 032065, Salta
  - Investigational Site Number 032051, San Miguel de Tucumán
  - Investigational Site Number 032008, San Miguel de Tucumán
  - Investigational Site Number 032033, San Nicolás
  - Investigational Site Number 032045, Santa Fe
  - Investigational Site Number 032035, Santa Fe
  - Investigational Site Number 032062, Santa Rosa
  - Investigational Site Number 032034, Venado Tuerto
  - Investigational Site Number 032046, Villa María
  - Investigational Site Number 032029, Zárate
- Australia (6):
  - Investigational Site Number 036015, Epping
  - Investigational Site Number 036001, Fremantle
  - Investigational Site Number 036009, Geelong
  - Investigational Site Number 036011, Perth
  - Investigational Site Number 036005, St Leonards
  - Investigational Site Number 036016, Townsville
- Austria (2):
  - Investigational Site Number 040002, Graz
  - Investigational Site Number 040001, Vienna
- Belarus (3):
  - Investigational Site Number 112002, Minsk
  - Investigational Site Number 112003, Minsk
  - Investigational Site Number 112001, Minsk
- Belgium (2):
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056003, Leuven
- Brazil (22):
  - Investigational Site Number 076024, Belém
  - Investigational Site Number 076006, Belo Horizonte
  - Investigational Site Number 076012, Belo Horizonte
  - Investigational Site Number 076021, Brasília
  - Investigational Site Number 076002, Campinas
  - Investigational Site Number 076019, Curitiba
  - Investigational Site Number 076003, Fortaleza
  - Investigational Site Number 076018, Fortaleza
  - Investigational Site Number 076004, Fortaleza
  - Investigational Site Number 076023, Goiânia
  - Investigational Site Number 076014, Marília
  - Investigational Site Number 076015, Passo Fundo
  - Investigational Site Number 076008, Porto Alegre
  - Investigational Site Number 076013, Porto Alegre
  - Investigational Site Number 076026, Porto Alegre
  - Investigational Site Number 076025, Recife
  - Investigational Site Number 076020, Salvador
  - Investigational Site Number 076016, São Paulo
  - Investigational Site Number 076010, São Paulo
  - Investigational Site Number 076001, São Paulo
  - Investigational Site Number 076005, São Paulo
  - Investigational Site Number 076007, Uberlândia
- Bulgaria (11):
  - Investigational Site Number 100002, Byala
  - Investigational Site Number 100011, Gabrovo
  - Investigational Site Number 100001, Kazanlak
  - Investigational Site Number 100006, Lovech
  - Investigational Site Number 100004, Pleven
  - Investigational Site Number 100003, Plovdiv
  - Investigational Site Number 100007, Plovdiv
  - Investigational Site Number 100016, Sandanski
  - Investigational Site Number 100010, Sofia
  - Investigational Site Number 100015, Sofia
  - Investigational Site Number 100005, Varna
- Canada (13):
  - Investigational Site Number 124024, Calgary
  - Investigational Site Number 124016, Cambridge
  - Investigational Site Number 124026, Edmonton
  - Investigational Site Number 124005, Greater Sudbury
  - Investigational Site Number 124001, Laval
  - Investigational Site Number 124021, Montreal
  - Investigational Site Number 124006, Montreal
  - Investigational Site Number 124027, Oshawa
  - Investigational Site Number 124025, Québec
  - Investigational Site Number 124028, Red Deer
  - Investigational Site Number 124003, Saint-Marc-des-Carrieres
  - Investigational Site Number 124007, Sarnia
  - Investigational Site Number 124002, Thetford-Mines
- Chile (29):
  - Investigational Site Number 152024, Antofagasta
  - Investigational Site Number 152023, Concepción
  - Investigational Site Number 152041, Osorno
  - Investigational Site Number 152040, Port Montt
  - Investigational Site Number 152038, Punta Arenas
  - Investigational Site Number 152036, San Felipe
  - Investigational Site Number 152035, Santiago
  - Investigational Site Number 152020, Santiago
  - Investigational Site Number 152028, Santiago
  - Investigational Site Number 152031, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152034, Santiago
  - Investigational Site Number 152008, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152019, Santiago
  - Investigational Site Number 152018, Santiago
  - Investigational Site Number 152042, Santiago
  - Investigational Site Number 152015, Santiago
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152029, Santiago
  - Investigational Site Number 152022, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152025, Talca
  - Investigational Site Number 152014, Temuco
  - Investigational Site Number 152003, Temuco
  - Investigational Site Number 152037, Valdivia
  - Investigational Site Number 152032, Valparaíso
  - Investigational Site Number 152010, Viña del Mar
  - Investigational Site Number 152002, Viña del Mar
- China (19):
  - Investigational Site Number 156016, Beijing
  - Investigational Site Number 156034, Beijing
  - Investigational Site Number 156024, Beijing
  - Investigational Site Number 156028, Beijing
  - Investigational Site Number 156014, Beijing
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156008, Dalian
  - Investigational Site Number 156020, Guangzhou
  - Investigational Site Number 156023, Jinan
  - Investigational Site Number 156015, Jinan
  - Investigational Site Number 156009, Nanjing
  - Investigational Site Number 156013, Shanghai
  - Investigational Site Number 156019, Shanghai
  - Investigational Site Number 156032, Shenyang
  - Investigational Site Number 156022, Shenyang
  - Investigational Site Number 156004, Suzhou
  - Investigational Site Number 156033, Ürümqi
- Colombia (19):
  - Investigational Site Number 170025, Armenia
  - Investigational Site Number 170009, Barranquilla
  - Investigational Site Number 170010, Barranquilla
  - Investigational Site Number 170002, Bogotá
  - Investigational Site Number 170005, Bogotá
  - Investigational Site Number 170012, Bogotá
  - Investigational Site Number 170014, Bogotá
  - Investigational Site Number 170022, Bogotá
  - Investigational Site Number 170004, Bucaramanga
  - Investigational Site Number 170017, Cali
  - Investigational Site Number 170024, Cali
  - Investigational Site Number 170013, Cartagena
  - Investigational Site Number 170026, Espinal - Tolima
  - Investigational Site Number 170007, Floridablanca
  - Investigational Site Number 170008, Floridablanca
  - Investigational Site Number 170019, Manizales
  - Investigational Site Number 170003, Medellín
  - Investigational Site Number 170020, Medellín
  - Investigational Site Number 170021, Pereira
- Denmark (11):
  - Investigational Site Number 208003, Aarhus
  - Investigational Site Number 208009, Aarhus C
  - Investigational Site Number 208011, Esbjerg
  - Investigational Site Number 208004, Farsø
  - Investigational Site Number 208002, Hellerup
  - Investigational Site Number 208010, Herlev
  - Investigational Site Number 208008, Hillerød
  - Investigational Site Number 208006, Hvidovre
  - Investigational Site Number 208001, København NV
  - Investigational Site Number 208005, København S
  - Investigational Site Number 208007, København Ø
- Ecuador (3):
  - Investigational Site Number 218001, Guayaquil
  - Investigational Site Number 218005, Guayaquil
  - Investigational Site Number 218002, Quito
- Egypt (2):
  - Investigational Site Number 818002, Alexandria
  - Investigational Site Number 818001, Cairo
- Estonia (6):
  - Investigational Site Number 233004, Tallinn
  - Investigational Site Number 233002, Tallinn
  - Investigational Site Number 233001, Tallinn
  - Investigational Site Number 233003, Tallinn
  - Investigational Site Number 233005, Tartu
  - Investigational Site Number 233006, Viljandimaa
- Finland (6):
  - Investigational Site Number 246005, Jyväskylä
  - Investigational Site Number 246003, Rauma
  - Investigational Site Number 246010, Tampere
  - Investigational Site Number 246009, Turku
  - Investigational Site Number 246007, Valkeakoski
  - Investigational Site Number 246012, Vantaa
- France (9):
  - Investigational Site Number 250008, Brest
  - Investigational Site Number 250002, Corbeil-Essonnes
  - Investigational Site Number 250005, Nantes
  - Investigational Site Number 250014, Nîmes
  - Investigational Site Number 250007, Paris
  - Investigational Site Number 250011, Pessac
  - Investigational Site Number 250012, Poitiers
  - Investigational Site Number 250006, Rennes
  - Investigational Site Number 250001, Toulouse
- Georgia (4):
  - Investigational Site Number 268003, Batumi
  - Investigational Site Number 268004, Kutaisi
  - Investigational Site Number 268001, Tbilisi
  - Investigational Site Number 268002, Tbilisi
- Germany (17):
  - Investigational Site Number 276003, Berlin
  - Investigational Site Number 276022, Bochum
  - Investigational Site Number 276005, Chemnitz
  - Investigational Site Number 276021, Dresden
  - Investigational Site Number 276024, Dresden
  - Investigational Site Number 276007, Elsterwerda
  - Investigational Site Number 276018, Frankfurt A.M.
  - Investigational Site Number 276011, Frankfurt am Main
  - Investigational Site Number 276017, Görlitz
  - Investigational Site Number 276025, Haßloch
  - Investigational Site Number 276009, Heidelberg
  - Investigational Site Number 276019, Leipzig
  - Investigational Site Number 276020, Magdeburg
  - Investigational Site Number 276028, Mühldorf
  - Investigational Site Number 276014, Pirna
  - Investigational Site Number 276016, Pohlheim
  - Investigational Site Number 276026, Rotenburg an der Fulda
- Guatemala (10):
  - Investigational Site Number 320004, Guatemala City
  - Investigational Site Number 320006, Guatemala City
  - Investigational Site Number 320012, Guatemala City
  - Investigational Site Number 320014, Guatemala City
  - Investigational Site Number 320001, Guatemala City
  - Investigational Site Number 320002, Guatemala City
  - Investigational Site Number 320007, Guatemala City
  - Investigational Site Number 320008, Guatemala City
  - Investigational Site Number 320011, Guatemala City
  - Investigational Site Number 320015, Quetzaltenango
- India (27):
  - Investigational Site Number 356019, Ahmedabad
  - Investigational Site Number 356002, Bangalore
  - Investigational Site Number 356010, Bangalore
  - Investigational Site Number 356026, Bangalore
  - Investigational Site Number 356024, Belagavi
  - Investigational Site Number 356012, Chandigarh
  - Investigational Site Number 356022, Gūrgaon
  - Investigational Site Number 356029, Hubli
  - Investigational Site Number 356020, Hyderabad
  - Investigational Site Number 356031, Jaipur
  - Investigational Site Number 356016, Kochi
  - Investigational Site Number 356004, Kolkata
  - Investigational Site Number 356015, Lucknow
  - Investigational Site Number 356014, Lucknow
  - Investigational Site Number 356009, Ludhiana
  - Investigational Site Number 356025, Madurai
  - Investigational Site Number 356032, Mangalore
  - Investigational Site Number 356018, Manipal
  - Investigational Site Number 356023, Mysore
  - Investigational Site Number 356027, Nagpur
  - Investigational Site Number 356006, Nagpur
  - Investigational Site Number 356030, Nashik
  - Investigational Site Number 356034, Nashik
  - Investigational Site Number 356013, New Delhi
  - Investigational Site Number 356017, New Delhi
  - Investigational Site Number 356021, Pune
  - Investigational Site Number 356028, Pune
- Israel (11):
  - Investigational Site Number 376010, Afula
  - Investigational Site Number 376006, Giv‘atayim
  - Investigational Site Number 376002, Haifa
  - Investigational Site Number 376008, Haifa
  - Investigational Site Number 376001, Holon
  - Investigational Site Number 376012, Jerusalem
  - Investigational Site Number 376011, Nahariya
  - Investigational Site Number 376005, Safed
  - Investigational Site Number 376004, Tel Aviv
  - Investigational Site Number 376003, Tel Litwinsky
  - Investigational Site Number 376009, Tzrifin
- Italy (16):
  - Investigational Site Number 380024, Carpi
  - Investigational Site Number 380004, Chieri
  - Investigational Site Number 380002, Chieti
  - Investigational Site Number 380006, Fermo
  - Investigational Site Number 380010, Florence
  - Investigational Site Number 380009, Genova
  - Investigational Site Number 380016, Messina
  - Investigational Site Number 380023, Milan
  - Investigational Site Number 380011, Milan
  - Investigational Site Number 380012, Milan
  - Investigational Site Number 380014, Napoli
  - Investigational Site Number 380019, Novara
  - Investigational Site Number 380005, Palermo
  - Investigational Site Number 380001, Pisa
  - Investigational Site Number 380013, Roma
  - Investigational Site Number 380020, Rozzano
- Japan (25):
  - Investigational Site Number 392011, Chūōku
  - Investigational Site Number 392015, Fuchu-Shi
  - Investigational Site Number 392012, Fujisawa-Shi
  - Investigational Site Number 392025, Hachioji-Shi
  - Investigational Site Number 392027, Hakusan-Shi
  - Investigational Site Number 392005, Hamamatsu
  - Investigational Site Number 392022, Hitachi-Shi
  - Investigational Site Number 392003, Itabashi-Ku
  - Investigational Site Number 392017, Itabashi-Ku
  - Investigational Site Number 392019, Kawanishi-Shi
  - Investigational Site Number 392013, Kobe
  - Investigational Site Number 392007, Matsuyama
  - Investigational Site Number 392008, Matsuyama
  - Investigational Site Number 392009, Nagasaki
  - Investigational Site Number 392002, Noda
  - Investigational Site Number 392020, Osaka
  - Investigational Site Number 392021, Osaka
  - Investigational Site Number 392001, Sapporo
  - Investigational Site Number 392010, Sapporo
  - Investigational Site Number 392024, Setagaya-Ku
  - Investigational Site Number 392004, Shinagawa-Ku
  - Investigational Site Number 392014, Shirakawa-Shi
  - Investigational Site Number 392018, Suita-Shi
  - Investigational Site Number 392016, Tachikawa-Shi
  - Investigational Site Number 392023, Takasaki-Shi
- Latvia (7):
  - Investigational Site Number 428005, Cēsis
  - Investigational Site Number 428001, Daugavpils
  - Investigational Site Number 428002, Liepāja
  - Investigational Site Number 428003, Riga
  - Investigational Site Number 428007, Riga
  - Investigational Site Number 428004, Riga
  - Investigational Site Number 428006, Sigulda
- Lithuania (6):
  - Investigational Site Number 440003, Kaunas
  - Investigational Site Number 440002, Kaunas
  - Investigational Site Number 440004, Klaipėda
  - Investigational Site Number 440006, Klaipėda
  - Investigational Site Number 440005, Panevezys
  - Investigational Site Number 440001, Vilnius
- Mexico (28):
  - Investigational Site Number 484011, Acapulco
  - Investigational Site Number 484008, Aguascalientes
  - Investigational Site Number 484033, Aguascalientes
  - Investigational Site Number 484016, Chihuahua City
  - Investigational Site Number 484023, Ciudad Madero
  - Investigational Site Number 484007, Durango
  - Investigational Site Number 484001, Durango
  - Investigational Site Number 484041, Durango
  - Investigational Site Number 484032, Guadalajara
  - Investigational Site Number 484034, Guadalajara
  - Investigational Site Number 484014, Guadalajara
  - Investigational Site Number 484028, Guadalajara
  - Investigational Site Number 484021, Guadalajara
  - Investigational Site Number 484006, Guadalajara
  - Investigational Site Number 484018, Guadalajara
  - Investigational Site Number 484024, León
  - Investigational Site Number 484026, Mexico City
  - Investigational Site Number 484022, Mexico City
  - Investigational Site Number 484013, Mexico City
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484025, Monterrey
  - Investigational Site Number 484002, Monterrey
  - Investigational Site Number 484005, Monterrey
  - Investigational Site Number 484004, Monterrey
  - Investigational Site Number 484035, Morelia
  - Investigational Site Number 484020, San Luis Potosí City
  - Investigational Site Number 484017, Tlalnepantla
  - Investigational Site Number 484031, Xalapa
- Netherlands (7):
  - Investigational Site Number 528005, Alkmaar
  - Investigational Site Number 528008, Deventer
  - Investigational Site Number 528004, Hoorn
  - Investigational Site Number 528001, Rotterdam
  - Investigational Site Number 528007, The Hague
  - Investigational Site Number 528003, Tilburg
  - Investigational Site Number 528006, Venlo
- Norway (3):
  - Investigational Site Number 578003, Bodø
  - Investigational Site Number 578002, Haugesund
  - Investigational Site Number 578001, Stavanger
- Panama (4):
  - Investigational Site Number 591001, Cuidad de Panama
  - Investigational Site Number 591003, Cuidad de Panama
  - Investigational Site Number 591004, La Chorrera
  - Investigational Site Number 591002, Penonomé
- Peru (15):
  - Investigational Site Number 604007, Arequipa
  - Investigational Site Number 604014, Callao
  - Investigational Site Number 604011, Lima
  - Investigational Site Number 604019, Lima
  - Investigational Site Number 604013, Lima
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604002, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604015, Lima
  - Investigational Site Number 604016, Lima
  - Investigational Site Number 604017, Lima
  - Investigational Site Number 604018, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604009, Lima
  - Investigational Site Number 604001, Lima
- Philippines (8):
  - Investigational Site Number 608006, Cavite
  - Investigational Site Number 608009, Iligan City, Lanao Del Norte
  - Investigational Site Number 608003, Makati City
  - Investigational Site Number 608001, Manila
  - Investigational Site Number 608007, Manila
  - Investigational Site Number 608005, Marikina City
  - Investigational Site Number 608002, Pasay
  - Investigational Site Number 608008, Quezon City
- Poland (20):
  - Investigational Site Number 616005, ?ód?
  - Investigational Site Number 616008, Bialystok
  - Investigational Site Number 616019, Bydgoszcz
  - Investigational Site Number 616012, Czeladź
  - Investigational Site Number 616007, Częstochowa
  - Investigational Site Number 616014, Gdynia
  - Investigational Site Number 616013, Gliwice
  - Investigational Site Number 616028, Grodzisk Mazowiecki
  - Investigational Site Number 616022, Katowice
  - Investigational Site Number 616001, Krakow
  - Investigational Site Number 616024, Krakow
  - Investigational Site Number 616023, Poland
  - Investigational Site Number 616021, Puławy
  - Investigational Site Number 616006, Ruda Śląska
  - Investigational Site Number 616025, Szczecin
  - Investigational Site Number 616032, Warsaw
  - Investigational Site Number 616020, Wroclaw
  - Investigational Site Number 616011, Wroclaw
  - Investigational Site Number 616031, Zgierz
  - Investigational Site Number 616029, Łęczyca
- Portugal (5):
  - Investigational Site Number 620005, Amadora
  - Investigational Site Number 620003, Coimbra
  - Investigational Site Number 620001, Lisbon
  - Investigational Site Number 620007, Penafiel
  - Investigational Site Number 620006, Porto
- Romania (22):
  - Investigational Site Number 642029, Arad
  - Investigational Site Number 642020, Baia Mare
  - Investigational Site Number 642003, Brasov
  - Investigational Site Number 642019, Brăila
  - Investigational Site Number 642034, Bucharest
  - Investigational Site Number 642022, Bucharest
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642013, Bucharest
  - Investigational Site Number 642026, Cluj-Napoca
  - Investigational Site Number 642030, Craiova
  - Investigational Site Number 642015, Craiova
  - Investigational Site Number 642007, Deva
  - Investigational Site Number 642011, Iași
  - Investigational Site Number 642010, Iași
  - Investigational Site Number 642016, Oradea
  - Investigational Site Number 642033, Piteşti
  - Investigational Site Number 642002, Ploieşti
  - Investigational Site Number 642009, Suceava
  - Investigational Site Number 642014, Târgu Mureş
  - Investigational Site Number 642012, Târgu Mureş
  - Investigational Site Number 642018, Timișoara
  - Investigational Site Number 642031, Timișoara
- Russia (55):
  - Investigational Site Number 643023, Barnaul
  - Investigational Site Number 643044, Kazan'
  - Investigational Site Number 643005, Kemerovo
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643061, Krasnodar
  - Investigational Site Number 643027, Krasnodar
  - Investigational Site Number 643037, Moscow
  - Investigational Site Number 643038, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643043, Moscow
  - Investigational Site Number 643008, Moscow
  - Investigational Site Number 643009, Moscow
  - Investigational Site Number 643029, Moscow
  - Investigational Site Number 643018, Moscow
  - Investigational Site Number 643042, Moscow
  - Investigational Site Number 643052, Moscow
  - Investigational Site Number 643026, Moscow
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643051, Moscow
  - Investigational Site Number 643013, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643060, Moscow
  - Investigational Site Number 643040, Moscow
  - Investigational Site Number 643034, Nizhny Novgorod
  - Investigational Site Number 643054, Novosibirsk
  - Investigational Site Number 643055, Novosibirsk
  - Investigational Site Number 643045, Omsk
  - Investigational Site Number 643030, Penza
  - Investigational Site Number 643017, Perm
  - Investigational Site Number 643049, Perm
  - Investigational Site Number 643048, Rostov-on-Don
  - Investigational Site Number 643047, Ryazan
  - Investigational Site Number 643024, Saint Petersburg
  - Investigational Site Number 643031, Saint Petersburg
  - Investigational Site Number 643035, Saint Petersburg
  - Investigational Site Number 643022, Saint Petersburg
  - Investigational Site Number 643039, Saint Petersburg
  - Investigational Site Number 643057, Saint Petersburg
  - Investigational Site Number 643041, Saint Petersburg
  - Investigational Site Number 643036, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643025, Saratov
  - Investigational Site Number 643056, Saratov
  - Investigational Site Number 643010, Saratov
  - Investigational Site Number 643033, Saratov
  - Investigational Site Number 643019, Saratov
  - Investigational Site Number 643014, Smolensk
  - Investigational Site Number 643028, Tomsk
  - Investigational Site Number 643016, Tver'
  - Investigational Site Number 643012, Tyumen
  - Investigational Site Number 643059, Vladimir
  - Investigational Site Number 643058, Voronezh
  - Investigational Site Number 643020, Yaroslavl
  - Investigational Site Number 643062, Yaroslavl
- Serbia (10):
  - Investigational Site Number 688002, Belgrade
  - Investigational Site Number 688003, Belgrade
  - Investigational Site Number 688004, Belgrade
  - Investigational Site Number 688006, Belgrade
  - Investigational Site Number 688008, Belgrade
  - Investigational Site Number 688009, Belgrade
  - Investigational Site Number 688010, Belgrade
  - Investigational Site Number 688001, Belgrade
  - Investigational Site Number 688005, Niš
  - Investigational Site Number 688007, Niš
- South Africa (16):
  - Investigational Site Number 710020, Alberton
  - Investigational Site Number 710017, Cape Town
  - Investigational Site Number 710006, Cape Town
  - Investigational Site Number 710010, Cape Town
  - Investigational Site Number 710025, Cape Town
  - Investigational Site Number 710008, Chatsworth
  - Investigational Site Number 710011, Durban
  - Investigational Site Number 710015, George
  - Investigational Site Number 710019, Kempton Park
  - Investigational Site Number 710014, Paarl
  - Investigational Site Number 710023, Parow
  - Investigational Site Number 710002, Pretoria
  - Investigational Site Number 710001, Pretoria
  - Investigational Site Number 710005, Richards Bay
  - Investigational Site Number 710007, Somerset West
  - Investigational Site Number 710004, Worcester
- South Korea (12):
  - Investigational Site Number 410012, Bucheon-si
  - Investigational Site Number 410006, Daegu
  - Investigational Site Number 410009, Gwangju
  - Investigational Site Number 410008, Incheon
  - Investigational Site Number 410001, Incheon
  - Investigational Site Number 410004, Seongnam
  - Investigational Site Number 410014, Seoul
  - Investigational Site Number 410013, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410011, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410007, Wŏnju
- Spain (15):
  - Investigational Site Number 724013, A Coruña
  - Investigational Site Number 724005, Alcalá de Henares
  - Investigational Site Number 724016, Almería
  - Investigational Site Number 724012, Barakaldo
  - Investigational Site Number 724018, Barcelona
  - Investigational Site Number 724014, Bilbao
  - Investigational Site Number 724015, Cáceres
  - Investigational Site Number 724008, Lleida
  - Investigational Site Number 724011, Madrid
  - Investigational Site Number 724017, Murcia
  - Investigational Site Number 724022, Oviedo
  - Investigational Site Number 724003, Pontevedra
  - Investigational Site Number 724001, Seville
  - Investigational Site Number 724020, Valencia
  - Investigational Site Number 724004, Vigo
- Sweden (7):
  - Investigational Site Number 752012, Karlstad
  - Investigational Site Number 752011, Kristianstad
  - Investigational Site Number 752006, Ljungby
  - Investigational Site Number 752009, Oskarshamn
  - Investigational Site Number 752004, Stockholm
  - Investigational Site Number 752007, Stockholm
  - Investigational Site Number 752002, Vaxjo
- Investigational Site Number 756003, Lugano, Switzerland
- Taiwan (8):
  - Investigational Site Number 158005, Chiayi City
  - Investigational Site Number 158004, Taichung
  - Investigational Site Number 158006, Tainan Hsien
  - Investigational Site Number 158002, Taipei
  - Investigational Site Number 158007, Taipei
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158008, Taipei
  - Investigational Site Number 158003, Taipei Hsien
- Tunisia (5):
  - Investigational Site Number 788003, Sfax
  - Investigational Site Number 788005, Tunis
  - Investigational Site Number 788004, Tunis
  - Investigational Site Number 788002, Tunis
  - Investigational Site Number 788001, Tunis
- Turkey (Türkiye) (11):
  - Investigational Site Number 792004, Ankara
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792012, Ankara
  - Investigational Site Number 792001, Capa / Istanbul
  - Investigational Site Number 792015, Istanbul
  - Investigational Site Number 792008, Istanbul
  - Investigational Site Number 792014, Istanbul
  - Investigational Site Number 792003, Izmir
  - Investigational Site Number 792007, Izmir
  - Investigational Site Number 792011, Mersin
  - Investigational Site Number 792013, Samsun
- Ukraine (12):
  - Investigational Site Number 804004, Chernivtsi
  - Investigational Site Number 804006, Dnipro
  - Investigational Site Number 804002, Dnipropetrovsk
  - Investigational Site Number 804009, Kharkiv
  - Investigational Site Number 804010, Kharkiv
  - Investigational Site Number 804003, Kiev
  - Investigational Site Number 804011, Kiev
  - Investigational Site Number 804012, Kyiv
  - Investigational Site Number 804013, Kyiv
  - Investigational Site Number 804005, Lviv
  - Investigational Site Number 804007, Odesa
  - Investigational Site Number 804008, Odesa
- United Arab Emirates (2):
  - Investigational Site Number 784001, Abu Dhabi
  - Investigational Site Number 784002, Dubai
- United Kingdom (31):
  - Investigational Site Number 826042, Antrim
  - Investigational Site Number 826002, Ashton-under-Lyne
  - Investigational Site Number 826026, Barnstaple
  - Investigational Site Number 826017, Bath
  - Investigational Site Number 826034, Birmingham
  - Investigational Site Number 826052, Bolton
  - Investigational Site Number 826005, Bradford
  - Investigational Site Number 826048, Carmarthen
  - Investigational Site Number 826037, Chester
  - Investigational Site Number 826011, Dumfries
  - Investigational Site Number 826044, East Kilbride
  - Investigational Site Number 826023, Edinburgh
  - Investigational Site Number 826008, Glasgow
  - Investigational Site Number 826010, Harrogate
  - Investigational Site Number 826040, Ipswich
  - Investigational Site Number 826033, Larbert
  - Investigational Site Number 826027, Liverpool
  - Investigational Site Number 826039, Londonderry
  - Investigational Site Number 826036, Manchester
  - Investigational Site Number 826021, Manchester
  - Investigational Site Number 826006, Manchester
  - Investigational Site Number 826049, Norwich
  - Investigational Site Number 826020, Nuneaton
  - Investigational Site Number 826009, Oldham
  - Investigational Site Number 826007, Salford
  - Investigational Site Number 826045, Stoke-on-Trent
  - Investigational Site Number 826038, Swansea
  - Investigational Site Number 826018, Taunton
  - Investigational Site Number 826016, Truro
  - Investigational Site Number 826046, Wolverhampton
  - Investigational Site Number 826019, Yeovil

REFERENCES:
- [Background] Bentley-Lewis R, Aguilar D, Riddle MC, Claggett B, Diaz R, Dickstein K, Gerstein HC, Johnston P, Kober LV, Lawson F, Lewis EF, Maggioni AP, McMurray JJ, Ping L, Probstfield JL, Solomon SD, Tardif JC, Wu Y, Pfeffer MA; ELIXA Investigators. Rationale, design, and baseline characteristics in Evaluation of LIXisenatide in Acute Coronary Syndrome, a long-term cardiovascular end point trial of lixisenatide versus placebo. Am Heart J. 2015 May;169(5):631-638.e7. doi: 10.1016/j.ahj.2015.02.002. Epub 2015 Feb 12. PMID 25965710
- [Result] Pfeffer MA, Claggett B, Diaz R, Dickstein K, Gerstein HC, Kober LV, Lawson FC, Ping L, Wei X, Lewis EF, Maggioni AP, McMurray JJ, Probstfield JL, Riddle MC, Solomon SD, Tardif JC; ELIXA Investigators. Lixisenatide in Patients with Type 2 Diabetes and Acute Coronary Syndrome. N Engl J Med. 2015 Dec 3;373(23):2247-57. doi: 10.1056/NEJMoa1509225. PMID 26630143
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Gerstein HC, Wolsk E, Claggett B, Diaz R, Dickstein K, Hess S, Kober L, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Tardif JC, Pfeffer MA. Effect of lixisenatide on natriuretic peptides in people with type 2 diabetes and recent acute coronary syndrome: The ELIXA trial. Diabetes Obes Metab. 2023 Apr;25(4):1125-1129. doi: 10.1111/dom.14954. Epub 2023 Jan 3. No abstract available. PMID 36546588
- [Derived] Gerstein HC, Hess S, Claggett B, Dickstein K, Kober L, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Tardif JC, Pfeffer MA. Protein Biomarkers and Cardiovascular Outcomes in People With Type 2 Diabetes and Acute Coronary Syndrome: The ELIXA Biomarker Study. Diabetes Care. 2022 Sep 1;45(9):2152-2155. doi: 10.2337/dc22-0453. PMID 35817031
- [Derived] Wijkman MO, Claggett B, Diaz R, Gerstein HC, Kober L, Lewis E, Maggioni AP, Wolsk E, Aguilar D, Bentley-Lewis R, McMurray JJ, Probstfield J, Riddle M, Tardif JC, Solomon SD, Pfeffer MA. Blood pressure and mortality in patients with type 2 diabetes and a recent coronary event in the ELIXA trial. Cardiovasc Diabetol. 2020 Oct 12;19(1):175. doi: 10.1186/s12933-020-01150-0. PMID 33046070
- [Derived] Shin SH, Claggett B, Pfeffer MA, Skali H, Liu J, Aguilar D, Diaz R, Dickstein K, Gerstein HC, Kober LV, Lawson FC, Lewis EF, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Tardif JC, Solomon SD; ELIXA Investigators. Hyperglycaemia, ejection fraction and the risk of heart failure or cardiovascular death in patients with type 2 diabetes and a recent acute coronary syndrome. Eur J Heart Fail. 2020 Jul;22(7):1133-1143. doi: 10.1002/ejhf.1790. Epub 2020 Mar 25. PMID 32212368
- [Derived] Seferovic JP, Bentley-Lewis R, Claggett B, Diaz R, Gerstein HC, Kober LV, Lawson FC, Lewis EF, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Solomon SD, Tardif JC, Pfeffer MA. Retinopathy, Neuropathy, and Subsequent Cardiovascular Events in Patients with Type 2 Diabetes and Acute Coronary Syndrome in the ELIXA: The Importance of Disease Duration. J Diabetes Res. 2018 Dec 16;2018:1631263. doi: 10.1155/2018/1631263. eCollection 2018. PMID 30648112
- [Derived] Muskiet MHA, Tonneijck L, Huang Y, Liu M, Saremi A, Heerspink HJL, van Raalte DH. Lixisenatide and renal outcomes in patients with type 2 diabetes and acute coronary syndrome: an exploratory analysis of the ELIXA randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2018 Nov;6(11):859-869. doi: 10.1016/S2213-8587(18)30268-7. Epub 2018 Oct 3. PMID 30292589
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361
- [Derived] Wolsk E, Claggett B, Pfeffer MA, Diaz R, Dickstein K, Gerstein HC, Lawson FC, Lewis EF, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Solomon SD, Tardif JC, Kober L. Role of B-Type Natriuretic Peptide and N-Terminal Prohormone BNP as Predictors of Cardiovascular Morbidity and Mortality in Patients With a Recent Coronary Event and Type 2 Diabetes Mellitus. J Am Heart Assoc. 2017 May 29;6(6):e004743. doi: 10.1161/JAHA.116.004743. PMID 28554908
- [Derived] Wohlfart P, Linz W, Hubschle T, Linz D, Huber J, Hess S, Crowther D, Werner U, Ruetten H. Cardioprotective effects of lixisenatide in rat myocardial ischemia-reperfusion injury studies. J Transl Med. 2013 Mar 28;11:84. doi: 10.1186/1479-5876-11-84. PMID 23537041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 829 centers in 49 countries. A total of 7719 participants were screened between June 24, 2010 and July 24, 2013. 1651 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: 7627 participants underwent 1 week placebo run-in period. 1559 were run-in failures due to exclusion criteria met. 6068 participants were randomized 1:1 to lixisenatide and placebo arms in double-blind treatment period. Duration of study was event driven until approximately 844 positively adjudicated primary cardiovascular (CV) outcome events.
Groups:
- Placebo: Placebo matched to lixisenatide once daily (QD) subcutaneously (SC) up to end of treatment (median exposure: 23 months).
- Lixisenatide: Lixisenatide 10 mcg QD SC for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to end of treatment (median exposure: 22 months).
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 3034 | 3034
Treated | 3032 | 3031
Completed | 2924 | 2929
Not Completed | 110 | 105
Not completed — Lost to Follow-up | 14 | 11
Not completed — Withdrawal by Subject | 83 | 88
Not completed — Site termination by sponsor | 13 | 5
Not completed — Other than specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo matched to lixisenatide QD SC up to end of treatment (median exposure: 23 months).
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 3034 | 3034 | 6068
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.6) | 59.9 (9.7) | 60.3 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 938 | 923 | 1861
  Male | 2096 | 2111 | 4207
Race [Number; unit: participants]
  Caucasian/White | 2318 | 2258 | 4576
  Black | 103 | 118 | 221
  Asian/Oriental | 367 | 404 | 771
  Other | 246 | 254 | 500
Ethnicity [Number; unit: participants]
  Hispanic | 903 | 865 | 1768
  Not Hispanic | 2131 | 2169 | 4300
Qualifying Acute Coronary Syndrome (ACS) event [Number; unit: participants]
  ST-segment elevation myocardial infarction (MI) | 1317 | 1349 | 2666
  Non ST-segment elevation MI | 1183 | 1165 | 2348
  Unstable angina | 528 | 514 | 1042
  Unclassified | 4 | 5 | 9
  Not qualifying ACS event | 2 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — N=3032, 3033
  kg/m^2 | 30.2 (5.79) | 30.12 (5.6) | 30.16 (5.69)
Body Weight [Mean (Standard Deviation); unit: kg] — N=3032, 3033
  kg | 85.06 (19.64) | 84.64 (19.21) | 84.85 (19.43)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — N=3033, 3034
  Percentage of HbA1c | 7.64 (1.28) | 7.72 (1.32) | 7.68 (1.30)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — N=3034, 3031
  years | 9.38 (8.32) | 9.2 (8.19) | 9.29 (8.25)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurence of Primary CV Event: CV Death, Non-Fatal MI, Non-Fatal Stroke or Hospitalization for Unstable Angina
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the onset of primary CV endpoint over time. Number of observed participants with endpoint events were reported. A CV event adjudication committee (CAC) reviewed and adjudicated, in a blinded fashion, all potential events.
Time Frame: From randomization up to the end of study (median follow-up of 25 months)
Population: Intent-to-treat (ITT) population defined as all randomized participants analyzed according to the treatment group allocated at randomization.
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 3034 | 3034
participants | 399 | 406
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; Analysis was performed using Cox proportional hazards model with treatment groups, and region (North America, South and Central America, Western Europe, Eastern Europe, Africa/Near East, and Asia/Pacific) as covariates, and the associated two-sided 95% confidence interval (CI); Test type: Non-Inferiority or Equivalence — Non-inferiority of lixisenatide versus placebo was to be claimed if the upper bound of the 2-sided 95% CI of the hazard ratio was <1.3; Hazard Ratio (HR) = 1.017, 95% CI 2-sided [0.886 to 1.168] — Lixisenatide vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Lixisenatide; Analysis was performed using Cox proportional hazards model with treatment groups, and region (North America, South and Central America, Western Europe, Eastern Europe, Africa/Near East, and Asia/Pacific) as covariates, and the associated two-sided 95% CI. Superiority of lixisenatide versus placebo was to be claimed if the upper bound of the 2-sided 95% CI of the hazard ratio was <1.0; Test type: Superiority or Other; p = 0.8542, Log Rank; Hazard Ratio (HR) = 1.017, 95% CI 2-sided [0.886 to 1.168] — Lixisenatide vs Placebo

2. Secondary Outcome: Time to First Occurence of CV Event: CV Death, Non-Fatal MI, Non-Fatal Stroke, Hospitalization for Unstable Angina or Hospitalization For Heart Failure
Description: All CV events were positively adjudicated by the CAC, used in the analysis of the composite CV endpoint comprised of CV death, non-fatal MI, non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure. Number of observed participants with endpoint events were reported.
Time Frame: From randomization up to the end of study (median follow-up of 25 months)
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 3034 | 3034
participants | 469 | 456

3. Secondary Outcome: Time to First Occurence of CV Event: CV Death, Non-Fatal MI, Non-Fatal Stroke, Hospitalization for Unstable Angina, Hospitalization For Heart Failure or Coronary Revascularization Procedure
Description: All CV events were positively adjudicated by CAC, used in the analysis of the composite CV endpoint comprised of CV death, non-fatal MI, non-fatal stroke, hospitalization for unstable angina, hospitalization for heart failure, or coronary revascularization procedure. Number of observed participants with endpoint events were reported.
Time Frame: From randomization up to the end of study (median follow-up of 25 months)
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 3034 | 3034
participants | 659 | 661

4. Secondary Outcome: Percent Change From Baseline in the Urinary Albumin/Creatinine Ratio (UACR) at Week 108
Description: Presence of albumin in urine is a marker of nephropathy, an important microvascular complication of diabetes. UACR was defined as the ratio: mg of albumin per gram of creatinine. UACR data were log transformed before the analysis. Calculation was based on geometric mean.
Time Frame: Baseline to Week 108 (LOCF)
Population: ITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline UACR value. Missing data was imputed using last observation carried forward (LOCF) using the last available post-baseline UACR before Week 108 as the value at Week 108, regardless of treatment discontinuation or not.
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 2830 | 2803
percent change | 34.21 (3.09) | 24.17 (2.84)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to study end (maximum follow-up of 52 months) regardless of seriousness or relationship to investigational medicinal product (IMP). Cardiovascular efficacy endpoint events were collected and analyzed separately within same time frame.
Description: Reported AEs are treatment emergent AEs that developed/worsened during 'on treatment period' (time from first administration of IMP up to 3 days after the last administration of IMP). Analysis was done on safety population that included all randomized participants received at least one dose of IMP.
Groups:
- Placebo: Participants exposed to Placebo matched to lixisenatide QD. (Median exposure: 23 months)
- Lixisenatide: Participants exposed to Lixisenatide 10 mcg QD SC for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to 225 weeks. (Median exposure: 22 months)
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 669/3032 | 625/3031
Other Adverse Events (participants affected / at risk) | 1270/3032 | 1597/3031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3032) | Lixisenatide (N=3031)
Pneumonia (Infections and infestations) | 51 | 36
Urinary tract infection (Infections and infestations) | 19 | 18
Cellulitis (Infections and infestations) | 18 | 17
Gastroenteritis (Infections and infestations) | 9 | 13
Sepsis (Infections and infestations) | 10 | 8
Bronchopneumonia (Infections and infestations) | 2 | 6
Respiratory tract infection (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 2 | 5
Osteomyelitis (Infections and infestations) | 9 | 4
Anal abscess (Infections and infestations) | 2 | 3
Appendicitis (Infections and infestations) | 3 | 3
Diverticulitis (Infections and infestations) | 1 | 3
Erysipelas (Infections and infestations) | 7 | 3
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Post procedural infection (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 5 | 3
Pyelonephritis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Abdominal sepsis (Infections and infestations) | 1 | 2
Diabetic foot infection (Infections and infestations) | 0 | 2
Empyema (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 7 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Infected skin ulcer (Infections and infestations) | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis chronic (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 3 | 2
Tooth abscess (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 2 | 2
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1
Gallbladder abscess (Infections and infestations) | 1 | 1
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 1
Infected bites (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 0 | 1
Mycobacterial infection (Infections and infestations) | 0 | 1
Nail bed infection (Infections and infestations) | 0 | 1
Osteomyelitis fungal (Infections and infestations) | 0 | 1
Paraspinal abscess (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Puncture site abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 4 | 1
Renal abscess (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 3 | 1
Toxoplasmosis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 3 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Burn infection (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Cat scratch disease (Infections and infestations) | 1 | 0
Chronic hepatitis B (Infections and infestations) | 1 | 0
Chronic hepatitis C (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 2 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Pleurisy viral (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Tick-borne fever (Infections and infestations) | 1 | 0
Viral corneal ulcer (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 10
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Iris melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 8
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 3
Drug hypersensitivity (Immune system disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 18 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Conversion disorder (Psychiatric disorders) | 1 | 0
Syncope (Nervous system disorders) | 16 | 16
Presyncope (Nervous system disorders) | 0 | 4
Carotid artery stenosis (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2
Hypoglycaemic unconsciousness (Nervous system disorders) | 3 | 2
Migraine (Nervous system disorders) | 0 | 2
Brain injury (Nervous system disorders) | 0 | 1
Carotid artery dissection (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 3 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 1
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Essential tremor (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 4 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Morton's neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 5 | 4
Cataract nuclear (Eye disorders) | 0 | 1
Diabetic retinal oedema (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 3 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Arteriosclerotic retinopathy (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Diabetic eye disease (Eye disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 3
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 23 | 23
Atrial fibrillation (Cardiac disorders) | 30 | 23
Ventricular tachycardia (Cardiac disorders) | 8 | 9
Coronary artery disease (Cardiac disorders) | 5 | 4
Atrial flutter (Cardiac disorders) | 5 | 3
Arrhythmia (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 8 | 2
Bradycardia (Cardiac disorders) | 5 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 3 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bifascicular block (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 5 | 1
Supraventricular tachycardia (Cardiac disorders) | 4 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 13 | 15
Deep vein thrombosis (Vascular disorders) | 2 | 5
Hypertension (Vascular disorders) | 9 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 5
Peripheral artery stenosis (Vascular disorders) | 2 | 5
Intermittent claudication (Vascular disorders) | 4 | 3
Aortic stenosis (Vascular disorders) | 2 | 2
Extremity necrosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 6 | 2
Leriche syndrome (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 4 | 2
Peripheral artery aneurysm (Vascular disorders) | 0 | 2
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial disorder (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 2 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 3 | 1
Peripheral vascular disorder (Vascular disorders) | 4 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 2 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 2 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 1 | 0
Vasculitis necrotising (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 4 | 7
Inguinal hernia (Gastrointestinal disorders) | 3 | 5
Duodenal ulcer (Gastrointestinal disorders) | 3 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 2
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 3 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 2 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faecal vomiting (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 2 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 3 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 6 | 13
Cholecystitis acute (Hepatobiliary disorders) | 7 | 10
Cholecystitis (Hepatobiliary disorders) | 5 | 9
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 | 8
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 20 | 20
Nephrolithiasis (Renal and urinary disorders) | 8 | 7
Renal failure (Renal and urinary disorders) | 5 | 6
Renal failure chronic (Renal and urinary disorders) | 4 | 6
Calculus urinary (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 5
Prostatitis (Reproductive system and breast disorders) | 1 | 2
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Vulval ulceration (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 42 | 46
Chest pain (General disorders) | 0 | 3
Death (General disorders) | 2 | 3
Coronary artery restenosis (General disorders) | 2 | 2
Arterial restenosis (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Multi-organ failure (General disorders) | 1 | 1
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Implant site extravasation (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 2
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose fluctuation (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 4 | 1
Blood pressure increased (Investigations) | 1 | 1
Carbohydrate antigen 19-9 increased (Investigations) | 0 | 1
Cardiac pacemaker evaluation (Investigations) | 0 | 1
Crystal urine present (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Angiogram (Investigations) | 1 | 0
Blood glucose abnormal (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 2 | 0
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 7
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 2 | 2
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 8 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Sports injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Cardioplegia (Surgical and medical procedures) | 0 | 1
Debridement (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 1
Pleurodesis (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 0
Intraocular lens implant (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Peripheral artery bypass (Surgical and medical procedures) | 1 | 0
Joint prosthesis user (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3032) | Lixisenatide (N=3031)
Nasopharyngitis (Infections and infestations) | 188 | 181
Hypoglycaemia (Metabolism and nutrition disorders) | 554 | 609
Dizziness (Nervous system disorders) | 191 | 259
Headache (Nervous system disorders) | 148 | 187
Angina pectoris (Cardiac disorders) | 200 | 177
Hypertension (Vascular disorders) | 171 | 152
Nausea (Gastrointestinal disorders) | 179 | 659
Vomiting (Gastrointestinal disorders) | 82 | 257
Diarrhoea (Gastrointestinal disorders) | 227 | 237
Non-cardiac chest pain (General disorders) | 171 | 137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.